CLINICAL TRIAL: NCT04343287
Title: A Multi-Center, Randomized, Double Masked, Placebo Controlled Clinical Study to Assess the Safety and Efficacy of BRM421 Ophthalmic Solution in Subjects With Dry Eye Using a Controlled Adverse Environment (CAE®) Model
Brief Title: Safety and Efficacy of BRM421 for Dry Eye Syndrome Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BRIM Biotechnology Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRM421-18-C001-PR
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Results first posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Masking
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BRM421 Ophthalmic Solution (Active Comparator): A topical solution of BRIM421 ophthalmic drops
  Interventions: Drug: BRM421
- Placebo (Placebo Comparator): A vehicle ophthalmic drops
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BRM421 — The active control with BRM421 solution
  Arms: BRM421 Ophthalmic Solution
Drug: Placebo — The vehicle solution
  Arms: Placebo

SUMMARY:
The objective of this study is to compare the safety and efficacy of BRM421 Ophthalmic Solution to placebo for the treatment of the signs and symptoms of dry eye.

DETAILED DESCRIPTION:
This is a multi-center, double-masked, randomized, placebo-controlled, phase 2/3 study with approximately 200 subjects. (around 100 subjects per treatment arm).

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Have a reported history of dry eye for at least 6 months prior to enrollment;
* Have a history of use of eye drops

Exclusion Criteria:

* Have any clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
* Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
* Have used any eye drops within 2 hours of Visit 1;
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
* Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Andover Eye Associates; Blair Boehmer, MD, Principal Investigator — Midwest Cornea Associates, LLC.; David Wirta, MD, Principal Investigator — Eye Research Foundation; Eugene B McLaurin, MD, Principal Investigator — Total Eye Care, PA
Locations (4):
- United States (4):
  - Eye Research Foundation, Newport Beach, California
  - Midwest Cornea Associates, LLC, Indianapolis, Indiana
  - Andover Eye Associates, Andover, Massachusetts
  - Total Eye Care, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BRM421 Ophthalmic Solution | Placebo
Started | 108 | 112
Completed | 108 | 111
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | BRM421 Ophthalmic Solution | Placebo | Total
Number analyzed (Participants) | 108 | 112 | 220
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 57 | 107
  >=65 years | 58 | 55 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (10.9) | 63.4 (12.07) | 63.7 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 83 | 152
  Male | 39 | 29 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 100 | 106 | 206
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 9 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 19 | 40
  White | 82 | 84 | 166
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 108 | 112 | 220
Total Corneal Fluorescein Staining (0-12: Higher is Worse) [Mean (Standard Deviation); unit: units on a scale] | 6.19 (0.904) | 6.15 (0.835) | 6.17 (0.868)
Dryness from Ocular Discomfort & 4-Symptom Questionnaire (0-5: Higher is Worse) [Mean (Standard Deviation); unit: units on a scale] | 3.0 (1.00) | 3.3 (0.93) | 3.2 (0.97)

OUTCOME MEASURES:

1. Primary Outcome: Ocular Sign: Change From Baseline in Total Corneal Staining Score to Day 14
Description: Corneal staining was performed to grade the degree of corneal epithelial cell injury as measured by fluorescence using slit-lamp examination. Ora Calibra® Scale from 0 to 4 with the use of half grade (0.5) increments, where grade 0 = None and 4 = Severe. Regions assessed were the central, superior, inferior, temporal, and nasal. Total corneal staining score was the sum of all five regions. Analyses were for study eye only.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BRM421 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 81 | 83
score on a scale | -1 (1.245) | -0.68 (1.392)

2. Primary Outcome: Ocular Symptom: Change From Baseline in Patient-Reported Ocular Dryness Score to Day 14, Using Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire
Description: Ocular dryness from the Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire was assessed at the subject level in regard to how both eyes felt. The Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire was used, which included rating the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging. Each symptom rating ranged from 0 to 5, where 0 = None and 5 = Worst.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BRM421 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 108 | 112
units on a scale | -0.3 (0.98) | -0.5 (0.99)

3. Secondary Outcome: Eye Dryness: Change From Baseline in Patient-Reported Ocular Symptom to Day 14, Using Visual Analog Scale (VAS)
Description: Visual analog scale (VAS) was measured by asking subjects to rate each ocular symptom due to ocular dryness by placing a vertical mark on a horizontal line of length 100 mm to indicate the level of discomfort where 0 mm = No Discomfort and 100 mm = Maximal Discomfort. Symptoms assessed were burning/stinging, itching, foreign body sensation, blurred vision, eye dryness, photophobia, and pain.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BRM421: The active control with BRM421 solution
  BRM421: A topical solution of BRIM421 ophthalmic drops
Arm/Group | BRM421 | Placebo
Number analyzed (Participants) | 108 | 112
score on a scale | -8.4 (19.22) | -3.7 (18.29)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | BRM421 Ophthalmic Solution | Placebo
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/112
Serious Adverse Events (participants affected / at risk) | 1/108 | 0/112
Other Adverse Events (participants affected / at risk) | 38/108 | 46/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BRM421 Ophthalmic Solution (N=108) | Placebo (N=112)
Osteomyelitis-left second toe/Infections and infestations/Osteomyelitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BRM421 Ophthalmic Solution (N=108) | Placebo (N=112)
instillation site pain (Eye disorders) | 38 | 46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT04343287/Prot_SAP_000.pdf